CLINICAL TRIAL: NCT05866289
Title: Awake Prone Positioning for COVID-19 Acute Hypoxaemic Respiratory Failure: Retrospective Cohort Study
Brief Title: Awake Prone Positioning for COVID-19 Acute Hypoxaemic Respiratory Failure
Status: Completed | Type: Observational
Sponsor: Mohammed VI University Hospital (Other)
Responsible Party: Principal Investigator, Younes Oujidi, Medical doctor, Mohammed VI University Hospital
Other Study IDs: unit critical care
Record Dates: First submitted 2023-03-27; First posted 2023-05-19 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Survival, Prosthesis; Oxygen Deficiency
Keywords: acute respiratory distress syndrome; COVID-19; conscious; prone position; survival rate
MeSH Terms: conditions — Prosthesis Failure; Hypoxia; Respiratory Distress Syndrome; COVID-19 | interventions — Prone Position

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 22 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Includes 681 patients who were placed in prone position
  Interventions: Other: Prone position
- Includes 388 patients who were placed in supine position

INTERVENTIONS:
Other: Prone position — Each prone position session had a minimum duration of one hour and a maximum duration of 12 hours for a minimum of 3 hours per day.
  Groups: Includes 681 patients who were placed in prone position

SUMMARY:
The objective of our study is to evaluate the effectiveness of prone position in preventing intubation or death in spontaneously ventilated patients with COVID-19 with acute respiratory failure.

DETAILED DESCRIPTION:
The COVID-19 pandemic has challenged the management of hypoxemic respiratory failure as limited ICU capacity is strained by a new high-mortality disease and large numbers of patients requiring prolonged periods of hospitalization, as well as respiratory support equipment such as ventilators and intensive care unit (ICU) beds.

If early and prolonged prone positioning (DV) reduces mortality in invasively ventilated patients with acute respiratory distress syndrome (ARDS), its role in conscious patients (DV vigil) remains a subject of debate and research.

This is a retrospective, monocentric, descriptive and analytical cohort conducted over a period of 22 months from March 2020 to December 2021 and involving 1069 patients hospitalized in the intensive care unit of the CHU Mohammed VI of Oujda for the management of acute respiratory failure caused by COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* all patients (1069 patients) with ARDS due to SARS-cov2, confirmed by nasopharyngeal swab, who were hospitalized in the COVID-19 ICU from March 1, 2020 to December 31, 2021

Exclusion Criteria:

* Patients with negative CRP
* Younger than 18 years of age
* Patients who died or intubated on the day of admission
* Patients presented a contraindication

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Each awake prone position session had a minimum duration of one hour and a maximum duration of 12 hours for a minimum of 3 hours per day.
  Epidemiological, clinical, paraclinical, therapeutic and evolutionary data were collected using a data processing form including the different variables collected in the patients' medical records. These data were then computerized and analyzed using IBM SPSS version 21 software.
  Qualitative variables were described as numbers and/or percentages, and quantitative variables as mean ± standard deviation, or as median with interquartile range for variables not having a normal distribution.
Sampling Method: Non-Probability Sample
Enrollment: 1069 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-12-28 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Evaluate the effectiveness of awake prone position in preventing intubation or death in spontaneously ventilated patients with COVID-19 with acute respiratory failure. | 22 months
  Evaluate the effectiveness of awake prone position in preventing intubation or death in spontaneously ventilated patients with COVID-19 with acute respiratory failure.

SECONDARY OUTCOMES:
length of stay in intensive care unit, length of time from hospitalization to death, length of time from hospitalization to intubation. | 22 months
  length of stay in intensive care unit, length of time from hospitalization to death, length of time from hospitalization to intubation.

CONTACTS AND LOCATIONS:
Locations (1):
- Amine Elmouhib, Oujda, Morocco

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Winearls S, Swingwood EL, Hardaker CL, Smith AM, Easton FM, Millington KJ, Hall RS, Smith A, Curtis KJ. Early conscious prone positioning in patients with COVID-19 receiving continuous positive airway pressure: a retrospective analysis. BMJ Open Respir Res. 2020 Sep;7(1):e000711. doi: 10.1136/bmjresp-2020-000711. PMID 32895247
- [Background] Sztajnbok J, Maselli-Schoueri JH, Cunha de Resende Brasil LM, Farias de Sousa L, Cordeiro CM, Sansao Borges LM, Malaque CMSA. Prone positioning to improve oxygenation and relieve respiratory symptoms in awake, spontaneously breathing non-intubated patients with COVID-19 pneumonia. Respir Med Case Rep. 2020;30:101096. doi: 10.1016/j.rmcr.2020.101096. Epub 2020 May 19. PMID 32455107
- [Background] Despres C, Brunin Y, Berthier F, Pili-Floury S, Besch G. Prone positioning combined with high-flow nasal or conventional oxygen therapy in severe Covid-19 patients. Crit Care. 2020 May 26;24(1):256. doi: 10.1186/s13054-020-03001-6. No abstract available. PMID 32456663
- [Background] Ding L, Wang L, Ma W, He H. Efficacy and safety of early prone positioning combined with HFNC or NIV in moderate to severe ARDS: a multi-center prospective cohort study. Crit Care. 2020 Jan 30;24(1):28. doi: 10.1186/s13054-020-2738-5. PMID 32000806
- [Background] Retucci M, Aliberti S, Ceruti C, Santambrogio M, Tammaro S, Cuccarini F, Carai C, Grasselli G, Oneta AM, Saderi L, Sotgiu G, Privitera E, Blasi F. Prone and Lateral Positioning in Spontaneously Breathing Patients With COVID-19 Pneumonia Undergoing Noninvasive Helmet CPAP Treatment. Chest. 2020 Dec;158(6):2431-2435. doi: 10.1016/j.chest.2020.07.006. Epub 2020 Jul 15. No abstract available. PMID 32679237
- [Background] Coppo A, Bellani G, Winterton D, Di Pierro M, Soria A, Faverio P, Cairo M, Mori S, Messinesi G, Contro E, Bonfanti P, Benini A, Valsecchi MG, Antolini L, Foti G. Feasibility and physiological effects of prone positioning in non-intubated patients with acute respiratory failure due to COVID-19 (PRON-COVID): a prospective cohort study. Lancet Respir Med. 2020 Aug;8(8):765-774. doi: 10.1016/S2213-2600(20)30268-X. Epub 2020 Jun 19. PMID 32569585

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-05-16): https://cdn.clinicaltrials.gov/large-docs/89/NCT05866289/Prot_SAP_ICF_000.pdf